CLINICAL TRIAL: NCT06160947
Title: Impact of Chiropractic Care on Opioid Use Among Adults With Chronic Non-Cancer Spinal Pain: A Pilot Cluster Randomized Controlled Trial (ACCESS-DC Pilot)
Brief Title: The Effect of Chiropractic Care on Opioid Use for Chronic Spinal Pain: A Feasibility Study
Acronym: ACCESS-DC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Surgical Methods Centre, McMaster University (Unknown); Michael G. DeGroote Institute for Pain Research and Care (Unknown); Ontario Chiropractic Association (Unknown); Alliance for Healthier Communities (Unknown); Michael G. DeGroote National Pain Centre (Unknown); Canadian Chiropractic Research Foundation (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Peter C Emary, DC, PhD, Postdoctoral fellow, Michael G. DeGroote National Pain Centre, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-2023
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Back Pain
Keywords: Clinical trials, randomized; Feasibility study; Analgesics, opioid; Chiropractic
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Cluster-randomized, 2-arm, data analyst-blinded feasibility trial
Who Masked: Investigator
Masking Description: Due to the nature of the intervention, it will not be possible to blind patients, study personnel, or clinicians to treatment allocation. However, data analysts and investigators responsible for interpreting results will be blinded to treatment allocation until all data have been analyzed and interpreted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Medical Care (Active Comparator): This group will consist of eligible, consenting, participants attending centers randomized to ongoing usual medical care.
  Interventions: Other: Usual Medical Care
- Usual Medical Care + Chiropractic Care (Experimental): This group will consist of eligible, consenting, participants attending centers randomized to ongoing usual medical care plus chiropractic care.
  Interventions: Other: Usual Medical Care + Chiropractic Care

INTERVENTIONS:
Other: Usual Medical Care — In both the intervention and control arms of the study, usual medical care will be defined as any and all medical care provided to patients with chronic non-cancer back or neck pain at a Canadian CHC, including: primary care provider consultation visits, prescription medication (e.g., muscle relaxants, anti-inflammatories, anti-depressants, opioid and non-opioid analgesics), referral for diagnostic testing (e.g., lab work, imaging) or specialist consultation, as well as other co-interventions (e.g., visits with nurses, dieticians, social workers, or physiotherapists) as determined by their PCP. PCPs will also engage study participants in a formal effort to reduce their opioid use within the framework of each CHC's current opioid-reduction practices.
  Arms: Usual Medical Care
Other: Usual Medical Care + Chiropractic Care — Treatment sessions may include high-velocity, low-amplitude spinal manipulative therapy, as well as any or all of the following: spinal mobilization, soft-tissue massage/trigger point therapy, education and reassurance (e.g., pain management, ergonomic and activities of daily living recommendations), and home advice (e.g., icing, spinal stretching, core muscle strengthening, and cardiovascular exercises). As part of the intervention, chiropractic clinicians will engage PCPs in a collaborative effort to support opioid tapering. Consistent with current clinical practice guidelines, participants will be provided up to a maximum of 18 chiropractic visits during the active care period, although participants may continue with treatment after the 12-week period (e.g., one visit, every 2-4 weeks) to manage episodes of exacerbation/flare-up.
  Arms: Usual Medical Care + Chiropractic Care

SUMMARY:
The investigators will conduct a pilot cluster randomized controlled trial (RCT) of chiropractic care added to usual medical care, versus usual medical care alone, for adult patients prescribed opioid therapy for chronic non-cancer spinal pain at four community health centers (CHCs) in Canada. These centers provide services to communities and vulnerable populations with high unemployment rates, multiple co-morbidities, and high rates of chronic musculoskeletal disorders that are commonly managed with prescription opioids.

The investigators hypothesize that a full-scale (definitive) cluster RCT on the impact of chiropractic care on prescription opioid use for chronic non-cancer spinal pain will be feasible within the Canadian CHC context.

DETAILED DESCRIPTION:
The investigators will conduct a cluster-randomized, 2-arm, data analyst-blinded feasibility RCT at four Canadian CHCs. The CHCs will be paired on clinical characteristics (e.g., size of patient roster, geographic location), and one center from each pair will be randomized to the intervention and control groups. At each of the four centers, the investigators will recruit adult patients with active opioid prescriptions for chronic non-cancer spinal pain (minimum dose of 50 mg morphine equivalents daily) who are not currently receiving chiropractic care and are interested in reducing their opioid dose. Each center (cluster) will be allocated to provide 26 weeks of usual medical care plus chiropractic care or usual medical care alone to enrolled participants. Random cluster allocation will be performed by an investigator blinded to the intervention group assignment. To further minimize the possibility of selection bias, clusters will be identified and recruited before randomization, and all eligible (and consenting) patients in each cluster will be included. The pilot trial will be coordinated by the Methods Centre within the Department of Surgery at McMaster University.

The primary aims of this study will be to: (1) estimate recruitment rates at the individual centers, (2) explore adherence to the study protocol, (3) investigate completeness of data collection, and (4) assess the ability to follow-up participants. The investigators will incorporate qualitative methods during the pilot trial (i.e., convergent, mixed methods experimental design) to complement the feasibility measures. The investigators will also collect preliminary data on the outcomes planned for a definitive trial: opioid use, pain, disability, bothersomeness, satisfaction, and quality of life at 6, 12, 18, and 26 weeks from enrolment.

ELIGIBILITY:
Inclusion Criteria:

Clusters

* CHC in Canada
* Roster of ≥ 3,500 patients
* One or more opioid-reducing strategies implemented as part of their standard medical services (e.g., chart audits, tracked performance metrics related to high dose prescribing)

Participants

* Adult patients (aged ≥ 18 years)
* Diagnosis of chronic non-cancer spinal pain (i.e., back or neck pain of ≥ 12 weeks' duration, not associated with cancer)
* Actively receiving one or more opioid prescriptions (minimum dose of 50 mg MED, dispensed over a period of at least 3 consecutive months)
* Interested in reducing their opioid dose
* Cognitive ability and language skills required to complete the outcome measures
* Provision of informed consent

Exclusion Criteria:

Clusters

• CHCs that employ chiropractors or have currently established chiropractic programs

Participants

* Individuals already receiving chiropractic care
* Opioid-naive (or < 90 consecutive days of opioid prescription) at baseline
* Total active opioid dosage of < 50 mg MED at baseline
* Actively receiving treatment for opioid use disorder (e.g., methadone, naloxone)
* Spinal neoplasms or other 'red flag' diagnoses (e.g., fractures, infections, inflammatory arthritis, or cauda equina syndrome)
* Anticipated problems with the participant being available for follow-up (e.g., incarceration, or planned incarceration)
* The participant is or may be enrolled in a competing trial
* Prior enrolment in the ACCESS-DC trial
* Other reason to exclude the participant, as approved by the Methods Centre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Participant Enrolment | From start of enrollment up to 26 weeks (or study end)
  Participant enrolment will be assessed by monitoring screening and enrolment metrics, including: 1) initiation of screening and recruitment at CHCs, 2) proportion of eligible patients approached for participation, 3) proportion of patients who provide informed consent, and 4) length of time required to enrol approximately six participants at each CHC. All outcome measures will be aggregated and interpreted via a "traffic light" approach (i.e., "green light" - proceed with RCT, "yellow light" - proceed with changes, "red light" - do not proceed unless changes are possible).
Treatment Allocation | Baseline, 6-, 12-, 18- and 26-week follow-up
  Feasibility of the treatment allocation will be assessed using the following metrics: 1) adherence to chiropractic care in addition to usual medical care allocation, and 2) adherence to usual medical care allocation. All outcome measures will be aggregated and interpreted via a "traffic light" approach (i.e., "green light" - proceed with RCT, "yellow light" - proceed with changes, "red light" - do not proceed unless changes are possible).
Refinement of Data Collection Methods | Baseline, 6-, 12-, 18- and 26-week follow-up
  To refine the data collection methods, the following metrics will be reviewed: 1) proportion of participants with missing data for the primary clinical outcome, and 2) proportion of case report forms with missing data for the participant-reported outcomes (BQ, Bothersomeness questionnaire, EQ-5D-5L, and patient satisfaction). All outcome measures will be aggregated and interpreted via a "traffic light" approach (i.e., "green light" - proceed with RCT, "yellow light" - proceed with changes, "red light" - do not proceed unless changes are possible).
Compliance with the Protocol | Baseline, 6-, 12-, 18- and 26-week follow-up
  The following outcomes will be used to assess compliance with the protocol: 1) participant compliance with scheduled appointments, 2) proportion of participants who complete each follow-up visit, 3) proportion of participants who withdraw consent to participate in the trial, and 4) proportion of participants who cannot be located. All outcomes will be aggregated and interpreted via a "traffic light" approach (i.e., "green light" - proceed with RCT, "yellow light" - proceed with changes, "red light" - do not proceed unless changes are possible).

SECONDARY OUTCOMES:
Daily Prescribed Opioid Dosage | Baseline, 6-, 12-, 18- and 26-week follow-up
  CHC information technology personnel will extract opioid prescription data from participants' individual electronic medical records to obtain the dose of chronic non-cancer spinal pain-related opioid prescriptions from baseline to 26-week follow-up. Opioid dosage will be measured in milligrams (mg) of morphine equivalents daily (MED). To calculate the MED for each prescribed opioid, the investigators will multiply the quantity x the mg per unit dispensed x drug-specific conversion factors.
Risk of Higher-Dose Opioid Prescriptions | Baseline, 6-, 12-, 18- and 26-week follow-up
  CHC information technology personnel will extract opioid prescription data from participants' individual electronic medical records to obtain the dose of chronic non-cancer spinal pain-related opioid prescriptions. Opioid dosage will be dichotomized as either high (e.g., ≥ 90 mg) MED or low (e.g., < 90 mg) MED at baseline and each follow-up interval. The threshold for opioid dose will be dependent on the central tendency of MED in the patient sample. A sensitivity analysis will also be conducted using a threshold of 50 mg MED.
Number of Opioid Prescriptions | Baseline, 6-, 12-, 18- and 26-week follow-up
  CHC information technology personnel will extract opioid prescription data from participants' individual electronic medical records to obtain the number and type of chronic non-cancer spinal pain-related opioid prescriptions (i.e., unique opioid fills and subsequent refills) over the entire course of follow-up, tabulated at the end of follow-up.
Level of Pain Intensity, and Physical and Emotional Functioning as measured by the Bournemouth Questionnaire (BQ) | Baseline, 6-, 12-, 18- and 26-week follow-up
  The BQ consists of 7 items (i.e., pain intensity, function in activities of daily living, function in social activities, anxiety, depression levels, fear avoidance behavior, and locus of control/self-efficacy), each scored from 0-10 ("0" = no disability, "10" = complete disability) for a total of 70. To optimize interpretability, the investigators will convert mean effects to risk differences using the anchor-based minimally important difference (MID) of the BQ established for chronic low back pain patients.
Level of Bothersomeness of Spinal Pain | Baseline, 6-, 12-, 18- and 26-week follow-up
  Self-rated level of bothersomeness on a 5-point Likert scale from "Not at all bothersome" to "Extremely bothersome".
Level of Patient Satisfaction | 6-, 12-, 18- and 26-week follow-up
  Self-rated satisfaction with care on a 5-point Likert scale from "Very satisfied" to "Very dissatisfied".
Quality of Life as measured by the EuroQol 5 Domain (EQ-5D) (5 Level Version) | Baseline, 6-, 12-, 18- and 26-week follow-up
  Self-rated health status measured on 5 domains (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on a 5-point Likert scale from "No problems" to "Extreme problems".

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Emary, DC, PhD, Principal Investigator — McMaster University; Jason W Busse, DC, PhD, Study Director — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting information will be made available from the Central Contact Person/Principal Investigator on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication